CLINICAL TRIAL: NCT04932434
Title: Psilocybin Therapy for Depression and Anxiety in Parkinson's Disease: a Pilot Study
Brief Title: Psilocybin Therapy for Depression and Anxiety in Parkinson's Disease
Acronym: PDP1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Joshua Woolley, MD, PhD (Other)
Responsible Party: Sponsor-Investigator, Joshua Woolley, MD, PhD, Associate Professor, University of California, San Francisco
Organization: University of California, San Francisco (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20-32641
Record Dates: First submitted 2021-05-05; First posted 2021-06-21 (Actual); Last update posted 2025-01-01 (Actual); Status verified 2024-12

CONDITIONS: Parkinson Disease; Depression; Anxiety
Keywords: Parkinson Disease; Depression; Anxiety; Psilocybin; Psilocybin therapy; Movement disorder
MeSH Terms: conditions — Parkinson Disease; Depression; Anxiety Disorders; Movement Disorders

STUDY DESIGN:
Intervention Model Description: Single Group Assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Psilocybin therapy (Experimental): Participants will receive one or two doses of psilocybin in a monitored setting approximately two weeks apart, with preparation sessions before and integration sessions after.
  Interventions: Drug: Psilocybin therapy

INTERVENTIONS:
Drug: Psilocybin therapy — * Psilocybin administration session 1: 10mg delivered orally with psychological support and monitoring
  * Psilocybin administration session 2: 25mg delivered orally with psychological support and monitoring
  Other Names: 4-phosphoryloxy-N,N-dimethyltryptamine

SUMMARY:
The purpose of this study is to determine the safety, tolerability, and feasibility of psilocybin therapy for depression and anxiety in people with Parkinson's disease.

DETAILED DESCRIPTION:
This is an open-label single-arm pilot study of oral psilocybin therapy for depression and anxiety in people with Parkinson's Disease (PD). The primary goal is to examine safety, tolerability, and feasibility of the intervention in this patient population. We will enroll people ages 40 to 75 with clinically diagnosed early stage Parkinson's Disease (Hoehn and Yahr Stage 1-3 during an "off" period), who meet DSM-5 criteria for a depressive or anxious disorder and meet all other inclusion and exclusion criteria at screening. After baseline assessments, participants will complete preparation sessions designed to provide information about the psilocybin experience and to build rapport/trust with the study team. Next, participants will complete a first psilocybin administration session, receiving a low-moderate dose of 10 mg oral psilocybin in a supervised setting with safety monitoring by a physician. Participants who do not experience significant adverse events during or following the session will complete a second psilocybin administration session approximately two weeks later. During the second psilocybin administration session, participants will receive a moderate-high dose of 25 mg oral. The second session will involve the same procedures and level of monitoring as the first. Participants will subsequently complete multiple follow-up sessions designed to assess PD and psychiatric symptoms as well as to provide support as they process their psilocybin experiences. Follow-up will continue to 3 months after the second psilocybin administration session. Primary endpoints will assess safety, tolerability, and feasibility of study procedures. Exploratory efficacy endpoints will assess changes in depressive symptoms, anxious symptoms, and related measures of function.

ELIGIBILITY:
Inclusion Criteria:

* Age 40 to 75
* Comfortable speaking and writing in English
* Clinically diagnosed early stage Parkinson's Disease (Hoehn and Yahr Stage 1-3 during an "off" period) who meet DSM-5 criteria for a depressive or anxious disorder and meet all other inclusion and exclusion criteria at screening
* Currently experiencing depression and/or anxiety (a formal diagnosis is not necessary)
* Able to attend all in-person visits at UCSF as well as virtual visits
* Have a care partner/support person available throughout the study
* Have an established primary care provider, neurologist, or psychiatrist

Exclusion Criteria:

* Psychotic symptoms involving loss of insight
* Significant cognitive impairment
* Regular use of medications that may have problematic interactions with psilocybin, including but not limited to dopamine agonists, MAO inhibitors, N-methyl-D-aspartate (NMDAR) antagonists, antipsychotics, and stimulants
* A health condition that makes this study unsafe or unfeasible, determined by study physicians

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2021-08-15 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Parkinson's Disease (PD) symptom severity | Baseline to 30 days following last drug dose
  Measured by Unified Parkinson's Disease Rating Scale (MDS-UPDRS)
Suicide Risk | Baseline to 30 days following last drug dose
  Measured by Columbia Suicide Severity Rating Scale (C-SSRS)
Psychotic symptoms | Baseline to 30 days following last drug dose
  Measured by Enhanced Scale for the Assessment of Positive Symptoms for Parkinson's Disease (eSAPS-PD)
Psychotic symptoms | Baseline to 30 days following last drug dose
  Measured by Psychosis and Hallucinations Questionnaire in Parkinson's Disease (PsycH-Q)
Cognitive Safety | Baseline to 30 days following last drug dose
  Measured by Cambridge Neuropsychological Test Automated Battery (CANTAB)
Caregiver/support person-reported distress | Baseline to 90 days following last drug dose
  Measured by Neuropsychiatric Inventory Caregiver Distress Questionnaire (NPI-Q)
Participant-reported subjective experience | Measured on each drug administration session day, following drug dose
  Measured by 5-Dimensional Altered States of Consciousness Rating Scale (5D-ASC)
Safety and tolerability of psilocybin therapy for depression and anxiety in people with PD | Baseline to 3 months following last drug dose
  Incidence, severity, and frequency of Adverse Events (AEs) including Treatment-Emergent AEs (TEAEs) and Serious AEs (SAEs)
Recruitment rate | Baseline to 3 months following last drug dose
  Measured by the number of participants entering the trial multiplied by the number of months of active recruitment time
Retention rate | Baseline to 3 months following last drug dose
  The number of participants completing all stages of the study will be presented as a percentage of the number of total number of participants recruited
Treatment Satisfaction of psilocybin therapy for depression and anxiety in people with PD | Baseline to 3 months following last drug dose
  Measured by the treatment satisfaction questionnaire
  * 5-item scale, plus three free response questions
  * items are ranked from 1-to-7, with higher scores representing better treatment satisfaction

OTHER OUTCOMES:
Effects of psilocybin therapy on depression in people with PD (exploratory) | Baseline to 3 months following last drug dose
  Measured by the Montgomery-Asberg Depression Rating Scale (MADRS)
  * Each item is scored on a on a scale of 0 to 6, with a total score of 0 to 60
  * Higher scores correspond to worse outcomes
Effects of psilocybin therapy on anxiety in people with PD (exploratory) | Baseline to 3 months following last drug dose
  Changes in anxiety assessed by the Hamilton Anxiety (HAM-A) Rating Scale
  * Each item is scored on a scale of 0 to 4 with a total score range of 0-56
  * Higher total scores correspond to worse outcomes
Cognitive Flexibility | Baseline to 30 days following last drug dose
  Measured by the Probabilistic Reversal Learning (PRL) task
Cognitive Flexibility | Baseline to 30 days following last drug dose
  Measured by the Cognitive Control and Flexibility Questionnaire
Transformational Experience | Baseline to 90 days following last drug dose
  Measured by the study-specific Transformational Experiences Questionnaire (TEQ)
Self-report changes to wellbeing | Baseline to 90 days following last drug dose
  Measured by the Quality of Life in Neurological Disorders
  * Each item is scored on a scale of 1 to 5
  * Higher total scores correspond to worse outcomes
Self-report changes to wellbeing | Baseline to 90 days following last drug dose
  Measured using the Patient-Reported Outcomes Measurement Information Systems
  * Each item is scored on a scale of 1 to 5
  * Lower total scores correspond to worse outcomes

CONTACTS AND LOCATIONS:
Overall Officials: Joshua Woolley, MD/PhD, Principal Investigator — University of California, San Francisco; Ellen Bradley, MD, Study Director — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] GBD 2016 Parkinson's Disease Collaborators. Global, regional, and national burden of Parkinson's disease, 1990-2016: a systematic analysis for the Global Burden of Disease Study 2016. Lancet Neurol. 2018 Nov;17(11):939-953. doi: 10.1016/S1474-4422(18)30295-3. Epub 2018 Oct 1. PMID 30287051
- [Background] Weintraub D, Burn DJ. Parkinson's disease: the quintessential neuropsychiatric disorder. Mov Disord. 2011 May;26(6):1022-31. doi: 10.1002/mds.23664. PMID 21626547
- [Background] Maillet A, Krack P, Lhommee E, Metereau E, Klinger H, Favre E, Le Bars D, Schmitt E, Bichon A, Pelissier P, Fraix V, Castrioto A, Sgambato-Faure V, Broussolle E, Tremblay L, Thobois S. The prominent role of serotonergic degeneration in apathy, anxiety and depression in de novo Parkinson's disease. Brain. 2016 Sep;139(Pt 9):2486-502. doi: 10.1093/brain/aww162. Epub 2016 Aug 17. PMID 27538418
- [Background] Schapira AHV, Chaudhuri KR, Jenner P. Non-motor features of Parkinson disease. Nat Rev Neurosci. 2017 Jul;18(7):435-450. doi: 10.1038/nrn.2017.62. Epub 2017 Jun 8. PMID 28592904
- [Background] Weintraub D, Moberg PJ, Duda JE, Katz IR, Stern MB. Effect of psychiatric and other nonmotor symptoms on disability in Parkinson's disease. J Am Geriatr Soc. 2004 May;52(5):784-8. doi: 10.1111/j.1532-5415.2004.52219.x. PMID 15086662
- [Background] Barone P, Antonini A, Colosimo C, Marconi R, Morgante L, Avarello TP, Bottacchi E, Cannas A, Ceravolo G, Ceravolo R, Cicarelli G, Gaglio RM, Giglia RM, Iemolo F, Manfredi M, Meco G, Nicoletti A, Pederzoli M, Petrone A, Pisani A, Pontieri FE, Quatrale R, Ramat S, Scala R, Volpe G, Zappulla S, Bentivoglio AR, Stocchi F, Trianni G, Dotto PD; PRIAMO study group. The PRIAMO study: A multicenter assessment of nonmotor symptoms and their impact on quality of life in Parkinson's disease. Mov Disord. 2009 Aug 15;24(11):1641-9. doi: 10.1002/mds.22643. PMID 19514014
- [Background] Ishihara L, Brayne C. A systematic review of depression and mental illness preceding Parkinson's disease. Acta Neurol Scand. 2006 Apr;113(4):211-20. doi: 10.1111/j.1600-0404.2006.00579.x. PMID 16542159